CLINICAL TRIAL: NCT00413244
Title: The Cardiac Benefit of Androgen Replacement in Hypogonadal Males With Coronary Artery Disease Following Successful Percutaneous Coronary Intervention (PCI).
Brief Title: The Cardiac Benefit of Testosterone Replacement in Men With Low Testosterone Levels With Coronary Artery Disease After Successful Intervention of the Blockage or Narrowed Heart Artery
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Collaborators: Abbott (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: GCO 06-1081
Record Dates: First submitted 2006-12-18; First posted 2006-12-19 (Estimated); Results first posted 2017-01-05 (Estimated); Last update posted 2017-01-05 (Estimated); Status verified 2016-11

CONDITIONS: Coronary Artery Disease
Keywords: Hypogonadal; coronary artery disease; percutaneous coronary intervention (PCI)
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Androgel treatment (Experimental): Androgel 5 grams
  Androgel treatment - subjects will be instructed to begin the study drug at 1 week post entry into the study and will continue to take the study drug for a total of 6 months. The study drug has to be applied to the skin once daily for 6 months.
  Interventions: Drug: AndroGel 5 Grams
- Placebo (Placebo Comparator): Placebo - will be instructed to begin the study drug at 1 week post entry into the study and will continue to take the study drug for a total of 6 months. The study drug has to be applied to the skin once daily for 6 months.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: AndroGel 5 Grams — Placebo (randomization will occur on a 2:1 drug to placebo). A total of 50 subjects will be randomized to receive Androgel 5 grams and 25 subjects will be randomized to receive placebo.
  Androgel treatment/Placebo (after the treatment arm is assigned, subjects will be instructed to begin the study drug at 1 week post entry into the study and will continue to take the study drug for a total of 6 months. The study drug has to be applied to the skin once daily for 6 months.
  Arms: Androgel treatment
Drug: Placebo — Placebo (randomization will occur on a 2:1 drug to placebo). A total of 50 subjects will be randomized to receive Androgel 5 grams and 25 subjects will be randomized to receive placebo.
  Androgel treatment/Placebo (after the treatment arm is assigned, subjects will be instructed to begin the study drug at 1 week post entry into the study and will continue to take the study drug for a total of 6 months. The study drug has to be applied to the skin once daily for 6 months.
  Arms: Placebo

SUMMARY:
The purpose of the study is to find out if giving the study drug, Androgel (testosterone) as a testosterone replacement help bring the testosterone to an acceptable level and to find out if it will help improve heart condition in males with coronary artery disease (CAD) following successful percutaneous coronary intervention.

DETAILED DESCRIPTION:
Males with coronary heart disease have lower serum levels of bioavailable testosterone than men of a similar age with normal coronary angiograms (English, European Heart Journal, 2000). Low plasma testosterone has been associated with known risk factors for CHD, including age, obesity, hyperinsulinemia, diabetes, and adverse lipid profile.

Testosterone has also been shown in numerous studies to be a vasodilator. Recently, testosterone replacement compared with placebo, in hypogonadal men was shown to improve time to ischemic threshold, assessed by treadmill exercise testing at 4 and 12 weeks (Malkin, Heart, 2000). Prior studies had also shown a beneficial effect on exercise-induced ischemia in men with CAD, but not exclusively hypogonadal men (Jaffe,Br Heart J 1977; Rosano, Circulation, 1999; English, Circulation, 2000). In addition, this proposed study would be the first study to assess if the anti-anginal effects persists long term.

This is a randomized, double-blind, placebo-controlled study to evaluate the safety and efficacy of testosterone supplementation in hypogonadal men with coronary artery disease following successful revascularization with percutaneous coronary intervention (PCI). Only those men who had successful coronary artery revascularization, and on stable cardiac medical regimen for the prior 4 weeks will be included. Eligible patients will then be randomized on a 2:1 basis with 50 subjects receiving 5 grams of AndroGel and 25 subjects receiving placebo gel.

The men in this study who demonstrate hypogonadism represent a novel population to demonstrate the safety and efficacy of testosterone supplementation to improve cardiac function and outcomes. We hypothesize that treatment of hypogonadism in men with CAD, following successful PCI, will significantly improve cardiac ischemic threshold as assessed by cardiac stress testing. Furthermore, additional cardiac endpoints such as angina status, endothelial function and inflammatory serum markers will also demonstrate significant benefit in the testosterone treated group.

ELIGIBILITY:
Inclusion Criteria:

* Adult male patients with coronary artery disease (CAD) (one to three vessel diseased).
* Stable cardiac status at least 3 months after percutaneous coronary intervention (PCI).
* No change in cardiac medications for 4 weeks prior to enrollment.
* Testosterone < 300 ng/dl or free testosterone < 5.0 ng/dl or bioavailable testosterone < 150 ng/dl.
* Sex Hormone Binding Globulin (SHBG) < 7nmol/liter and Free Testosterone < 50pg/dl
* Prostate Specific Antigen (PSA) < 2.5 ng/mL or 2.6-3.7ng/mL with a negative prostate biopsy within the last 6 months and pathology report available for investigator's review.
* Subgroup of diabetics with well to moderately controlled diabetes (defined by a HgbA1c of < 9mg/dL.

Exclusion Criteria:

* Hematocrit greater than 50%.
* Severe hypertension (exhibit systolic blood pressure >180mmHg and diastolic blood pressure >110 mmHg at baseline visit or a have a history of malignant hypertension.
* Significant cardiac arrhythmia (supraventricular tachycardia [SVT] or ventricular tachycardia with heart rate exceeding 110 beats per minute at Visit 1).
* ECG abnormalities precluding ST segment analysis on treadmill, or inability to walk on treadmill.
* Poorly controlled, symptomatic, active medical problems (HIV, hepatitis, cancer, benign prostatic hypertrophy, alcohol or drug abuse, major depressive disorder).
* Neurological or psychiatric disorder that would compromise the patient's ability to give informed consent or adhere to the requirements of the protocol.
* History of prostate cancer
* History of hypersensitivity to transdermal testosterone gel.
* International Prostate Symptom Score (IPSS) >19 at Visit 1.

Ages: 40 Years to 75 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2007-01; Primary Completion 2014-01 (Actual); Study Completion 2014-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mary Ann McLaughlin, MD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Icahn School of Medicine at Mount Sinai, New York, New York, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects recruited for the study were male patients with stable cardiac status at least 3 months after Percutaneous Coronary Intervention (PCI) at the Cardiac Catheterization Lab of Mount Sinai Hospital from July 2007 to August 2013.
Groups:
- Androgel: Androgel 5 grams
- Placebo: Matching Placebo
Period: Overall Study
Arm/Group | Androgel | Placebo
Started | 31 | 20
Completed | 21 | 19
Not Completed | 10 | 1
Not completed — Withdrawal by Subject | 10 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Androgel | Placebo | Total
Number analyzed (Participants) | 31 | 20 | 51
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.3 (8.2) | 58.9 (7.3) | 58.5 (7.81)
Gender [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 31 | 20 | 51
Hypertension [Number; unit: participants]
  Yes | 30 | 16 | 46
  No | 1 | 4 | 5
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] | 30.8 (5.8) | 28.0 (4.3) | 29.7 (5.4)
Diabetes [Number; unit: participants]
  Yes | 16 | 6 | 22
  No | 15 | 14 | 29
Total Testosterone [Mean (Standard Deviation); unit: ng/dL] | 246.7 (63.5) | 263.7 (71.9) | 253.36 (66.8)
Systolic Blood Pressure [Mean (Standard Deviation); unit: mmHg] | 123.81 (13.81) | 128.05 (20.84) | 125.47 (16.85)
Diastolic Blood Pressure [Mean (Standard Deviation); unit: mmHg] | 76.32 (9.03) | 75.10 (11.65) | 75.84 (10.04)
Hematocrit [Mean (Standard Deviation); unit: percent of cells] | 40.69 (3.00) | 40.93 (3.18) | 40.78 (3.04)
White Blood Cell Count [Mean (Standard Deviation); unit: cells x10^3/uL] | 6.25 (1.78) | 6.49 (1.63) | 6.34 (1.71)
Red Blood Cell Count [Mean (Standard Deviation); unit: cells x10^6/uL] | 4.58 (0.44) | 4.67 (0.42) | 4.62 (0.43)
Aging male syndrome questionnaire [Mean (Standard Deviation); unit: units on a scale] — The scale assesses symptoms of aging and their impact on HRQoL in males, and increases with increasing severity (1 to 5) of subjectively perceived complaints in 17 items. Scale ranges from 17-85 (no symptoms to extremely severe symptoms.)
  units on a scale | 36.48 (11.36) | 35.85 (10.24) | 36.24 (10.83)
Exercise Time [Mean (Standard Deviation); unit: seconds] | 507.29 (153.48) | 530.00 (120.08) | 516.20 (104.49)
International Prostate Symptom Score (IPSS) [Mean (Standard Deviation); unit: units on a scale] — IPSS has 8 questions total - 7 questions related to symptoms, each item scored 1-5. (asymptomatic to very symptomatic). The 8th question refers to the patient's perceived quality of life ranged from 0 to 6 ("delighted" to "terrible".) Total scale ranges from 8-35. Mild (symptom score less than of equal to 7) Moderate (symptom score range 8-19) Severe (symptom score range 20-35)
  units on a scale | 5.68 (4.77) | 4.55 (4.7) | 5.24 (4.73)
Metabolic equivalent of task (METs) [Mean (Standard Deviation); unit: MET units] | 10.03 (2.58) | 10.05 (1.99) | 10.04 (2.34)
Reactive hyperemia index (RHI) [Mean (Standard Deviation); unit: ml] | 1.97 (0.72) | 1.85 (0.54) | 1.92 (0.66)
Total Cholesterol [Mean (Standard Deviation); unit: mg/dL] | 157.29 (47.10) | 144.45 (28.85) | 152.25 (41.08)
LDL [Mean (Standard Deviation); unit: mg/dL] | 86.48 (40.52) | 80.90 (26.77) | 84.29 (35.57)
Triglycerides [Mean (Standard Deviation); unit: mg/dL] | 142.23 (100.95) | 109.90 (50.86) | 129.55 (85.74)
Waist Circumference [Mean (Standard Deviation); unit: inches] | 42.66 (5.21) | 41.31 (4.65) | 42.13 (4.99)
Weight [Mean (Standard Deviation); unit: lbs] | 205.73 (39.22) | 194.50 (36.62) | 201.32 (38.25)

OUTCOME MEASURES:

1. Primary Outcome: Cardiac Stress Test: Time to ST Depression
Description: Treadmill exercise testing performed according to the Bruce protocol (MAX-1 Marquette advanced exercise system, software version 002E). The system analyzed the signal averaged ECG and produces a graphical display of the level of the ST segment 80 ms after the J point against time. Time to 1 mm ST depression was measured from computer derived analysis, effectively eliminating observer bias.
Time Frame: at 6 months
Population: Subjects analyzed were only those subjects with ST depression at baseline
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Androgel | Placebo
Number analyzed (Participants) | 10 | 11
seconds
  at 1 month | 439.1 (205.2) | 279.5 (130.0)
  at 3 months | 364.0 (141.4) | 292.6 (63.5)
  at 6 months | 433.0 (123.2) | 342.2 (62.7)
Statistical Analysis 1: Comparison: Androgel vs Placebo; Statistician used all the time points post-baseline together ("Overall"). The result gives the estimates and 95% CI of the treatment effect from longitudinal analyses (generalized estimating equation method) which basically pools data from all visits post-baseline; Test type: Superiority or Other; p = 0.03, log mean

2. Primary Outcome: Cardiac Stress Testing: Exercise Capacity
Description: Exercise capacity was measured using exercise time.
Time Frame: At 1 month, 3 months, and 6 months
Population: Subjects analyzed were only those subjects with ST depression at baseline
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Androgel | Placebo
Number analyzed (Participants) | 10 | 11
seconds
  at 1 month | 589.7 (114.6) | 452.4 (122.7)
  at 3 months | 607.6 (152.0) | 472.1 (98.6)
  at 6 months | 614.0 (115.4) | 470.0 (143.8)

3. Secondary Outcome: Seattle Angina Questionnaire (SAQ)
Description: A cardiac disease-related quality-of-life measure. The SAQ is a self-report instrument with 19 items that, yields five subscale scores: physical limitation, angina stability, angina frequency, treatment satisfaction, and disease perception. The possible range of scores for each of the five subscales is 0 to 100, with higher scores indicating better quality of life. A change of 10 points in any of the subscales is considered to be clinically important.
  Data not collected.
Time Frame: up to 6 months
Arm/Group | Androgel | Placebo
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Reactive Hyperemia Index
Description: The Reactive Hyperemia Index measures the endothelial function and predicts future coronary events. In general RHI values below 2 are categorized as endothelial dysfunction and have a greater plaque burden, whereas higher RHI values are considered normal or improved endothelial function. PAT is the technique to non-invasively assess endothelial function. It comprises finger probes to evaluate digital volume changes.
Time Frame: 6 months
Population: Subjects analyzed were only those subjects with ST depression at baseline
Measure: Mean (Standard Deviation); unit: mls
Arm/Group | Androgel | Placebo
Number analyzed (Participants) | 10 | 11
mls
  At baseline | 1.96 (0.72) | 1.85 (0.54)
  at 1 month | 1.85 (0.49) | 1.81 (0.52)
  at 3 months | 1.70 (0.49) | 1.77 (0.37)
  at 6 moths | 1.83 (0.58) | 1.74 (0.53)

5. Secondary Outcome: International Prostate Symptom Score (IPSS)
Description: IPSS has 7 questions related to symptoms, each item scored 1-5. Total score can range from 0 to 35 (asymptomatic to very symptomatic). The 8th question refers to the patient's perceived quality of life ranged from 0 to 6 ("delighted" to "terrible".) Data not collected.
Time Frame: 6 months
Arm/Group | Androgel | Placebo
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Metabolic Equivalents of Task (METS)
Description: The Metabolic Equivalent of Task (MET), or simply metabolic equivalent, is a physiological measure expressing the energy cost of physical activities and is defined as the ratio of metabolic rate (and therefore the rate of energy consumption) during a specific physical activity to a reference metabolic rate, set by convention to 3.5 ml O2·kg-1·min-1 or equivalently
Time Frame: 6 months
Population: Subjects analyzed were only those subjects with ST depression at baseline
Measure: Mean (Standard Deviation); unit: METS units
Arm/Group | Androgel | Placebo
Number analyzed (Participants) | 10 | 11
METS units
  at baseline | 11.0 (2.2) | 9.0 (1.3)
  at 1 month | 11.4 (2.2) | 9.0 (1.9)
  at 3 months | 11.9 (3.0) | 9.2 (1.5)
  at 6 months | 12.2 (2.2) | 9.4 (2.3)

7. Secondary Outcome: Aging Male Symptoms (AMS)
Description: The scale assesses symptoms of aging and their impact on HRQoL in males, and increases with increasing severity (1 to 5) of subjectively perceived complaints in 17 items. Scale ranges from 17-85 (no symptoms to extremely severe symptoms.)
Time Frame: At baseline, 1 month, 3 months, and 6 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Androgel | Placebo
Number analyzed (Participants) | 31 | 20
units on a scale
  Baseline | 36.5 (11.4) | 35.8 (10.2)
  At 1 month | 32.9 (10.1) | 29.8 (11.6)
  At 3 months | 36.5 (11.4) | 35.9 (10.2)
  At 6 months | 31.2 (8.5) | 31.4 (9.8)

8. Secondary Outcome: International Index of Erectile Function (IIEF)
Description: Questions 1-5 15 of the IIEF relates to erectile function scale 0 - 30 (severe erectile dysfunction to no erectile dysfunction).
Time Frame: At baseline, 1 month, 3 months, and 6 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Androgel | Placebo
Number analyzed (Participants) | 31 | 20
units on a scale
  at baseline | 12.4 (8.7) | 12.2 (9.4)
  at 1 month | 14.1 (9.0) | 10.1 (9.2)
  at 3 months | 15.7 (9.6) | 14.2 (10.8)
  at 6 months | 15.0 (10.0) | 12.5 (9.7)

9. Secondary Outcome: IIEF-II Orgasmic Function
Description: Questions 9-10 of the IIEF relates to orgasmic function scale 0 - 10 (from no impairment to severe impairment)
Time Frame: At baseline, 1 month, 3 months, and 6 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Androgel | Placebo
Number analyzed (Participants) | 31 | 20
units on a scale
  at baseline | 4.8 (3.3) | 4.4 (3.6)
  at 1 month | 5.9 (3.5) | 4.2 (4.2)
  at 3 months | 5.7 (3.7) | 5.8 (4.2)
  at 6 months | 6.1 (3.4) | 5.5 (4.3)

10. Secondary Outcome: IIEF -III: Sexual Desire
Description: Questions 11-12 of the IIEF relates to sexual desire scale 0-10 (from very low to very high)
Time Frame: At baseline, 1 month, 3 months, and 6 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Androgel | Placebo
Number analyzed (Participants) | 31 | 20
units on a scale
  at baseline | 5.0 (2.1) | 5.4 (1.8)
  at 1 month | 5.6 (2.7) | 4.8 (2.4)
  at 3 months | 6.3 (2.3) | 5.6 (2.0)
  at 6 months | 6.6 (2.4) | 5.5 (2.6)

11. Secondary Outcome: IIEF-IV: Intercourse Satisfaction
Description: Questions 6,7, 8 of the IIEF relates to intercourse satisfaction scale 0 - 15 (from very dissatisfied to very satisfied)
Time Frame: At baseline, 1 month, 3 months, and 6 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Androgel | Placebo
Number analyzed (Participants) | 31 | 20
units on a scale
  at baseline | 5.5 (4.0) | 5.0 (4.6)
  at 1 month | 6.2 (4.6) | 3.6 (4.4)
  at 3 months | 6.8 (4.9) | 6.0 (5.1)
  at 6 months | 6.9 (5.1) | 5.2 (5.1)

12. Secondary Outcome: IIEF-V: Over-all Satisfaction
Description: Questions 13,14 of the IIEF relates to specifically to overall satisfaction scale from 0 - 10 (very dissatisfied to very satisfied)
Time Frame: At baseline, 1 month, 3 months, and 6 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Androgel | Placebo
Number analyzed (Participants) | 31 | 20
units on a scale
  at baseline | 4.8 (2.5) | 4.3 (2.4)
  at 1 month | 4.9 (2.9) | 3.8 (2.7)
  at 3 months | 5.2 (2.9) | 5.2 (3.0)
  at 6 months | 6.0 (3.0) | 4.9 (3.2)

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Androgel | Placebo
Serious Adverse Events (participants affected / at risk) | 0/31 | 0/20
Other Adverse Events (participants affected / at risk) | 0/31 | 0/20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes